CLINICAL TRIAL: NCT01547624
Title: Neck Muscle Activation in Patients With Long Standing Problems After a Whiplash Trauma Registered With Ultrasound With Speckle Tracking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anneli Peolsson, Assoc. Prof., PhD, MSC PT, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Ultrasound on neck muscles WAD
Record Dates: First submitted 2012-02-28; First posted 2012-03-08 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Whiplash Associated Disorder
Keywords: Neck; Spine; Muscles; Activity; Coordination
MeSH Terms: conditions — Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neck Specific exercises (Experimental): 3 months of neck specific exercises for 30 patients.
  Interventions: Other: Neck specific exercises
- Waiting list (No Intervention): Thirty patients on the waiting list for 3 month before they have their intervention
- Healthy controls (No Intervention): Forty healthy controls. Comparisons between forty included WAD patients and 40 healthy controls matched for age and gender will be investigated at baseline.

INTERVENTIONS:
Other: Neck specific exercises — Neck specific exercises 2 times/week for 3 month at a physiotherapist. Home exercises.
  Other Names: Physiotherapy with neck specific exercises
  Arms: Neck Specific exercises

SUMMARY:
Today there is evidence for that neck specific exercises reduce neck pain problems in patients with mechanical neck pain. However, there is a lack of consensus on how to optimize neck exercises and dosages in neck rehabilitation. More knowledge is needed to determine which and how muscles are activated in exercises thought to be neck-specific. There is neither enough knowledge of differences in neck muscle activation between patients with long standing neck problems after a whiplash trauma and healthy controls nor if the neck muscle function improved with specific neck exercises. One approach would be a real time study of deformation and deformation rate in different layers of neck muscles in patients with residual long-term neck pain and disability after a whiplash trauma. The purpose of the present study was to investigate deformation and deformation rate in different layers of dorsal and ventral neck muscles (including upper and middle part of trapezius muscle) during rest and during different exercises; arm flexion until 120 degrees, repeated arm flexion until 90 degrees, low loaded neck extension, low loaded neck muscle endurance test, shoulder elevation. Forty patients with long standing (more than 6 months but less than 3 years)patients and 40 controls matched for age and gender will be included for comparisons between patients and healthy in neck muscle activation. The investigators also include 60 patients with whiplash trauma, of those 30 patients will be randomized to A. neck specific exercises in a 3 months period and B. will 30 be on a waiting list for 3 months. Measurements are performed at baseline and at 3 months follow-up. Those patients who fulfilled the 3 months period of neck specific exercises will also be asked for a 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* WAD II and III
* Age 18-63 years
* Remaining problems
* Right handed
* Pain on right or on both sides.

Exclusion Criteria:

* Myelopathy
* Earlier fracture or luxation of the cervical column, earlier neck injury
* Spinal tumour
* Spinal infection
* Surgery in the cervical column
* Malignity
* Systemic disease or other disease or another injury contraindicated to perform the treatment program or the measurements
* Diagnosed severe psychiatric disorder
* Unconscious in connection to the trauma
* Known drug abuse
* Lack of familiarity with the Swedish language

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Speckle tracking analysis of muscle function | Baseline and at 3 and 6 months follow-up. The outcome measure is going to report a change over time.
  Measured with medical ultrasonography

SECONDARY OUTCOMES:
Background data | Baseline
  Background data of age, gender, social situation, work, work situation, sick-leave, income, pain history, debute of symptoms, about the accident, earlier treatment, other diseases or pain problems, expectations of treatment
Symptom satisfaction | Baseline and at 3 months follow-up. The outcome measure is going to report a change over time.
Pain intensity on visual analogue scale (VAS) | Baseline and at 3 months follow-up. The outcome measure is going to report a change over time.
  Symptoms in general, Neck, Arm, Headache
Dizziness/ unsteadiness on visual analogue scale | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
Pain distribution on drawing | Baseline and at 3 months follow-up. The outcome measure is going to report a change over time.
Pain Disability Index | Baseline and at 3 months follow-up. The outcome measure is going to report a change over time
Neck Disability Index | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
Tampa Scale of Kinesiophobia (TSK-11 short version) | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
Pain Catastrophizing Scale | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
Hospital Anxiety and Depression Scale | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
Euroquol | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
  Euroquol 5D and thermometer
Exercise Self-Efficacy Scale | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
  "How confident you are to exercise when things get in the way" Exercise self-efficacy scale is a six item scale with a five point scale (1=not at all confident and 5=completely confident).
Self-Efficacy Scale | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
  "People´s beliefs about their capabilities to produce designated levels of performance that exercise influence over events that affect their lives" Self-efficacy scale (by Altmaier) is a 20 item, 11 point scale (0=not at all confident, 10=completely confident).
Work Ability Index | Baseline and at 3 month follow-up. The outcome is going to report a change over time.
Physical Activity level | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.
Physical Outcome Measures | Baseline and at 3 month follow-up. The outcome is going to report a change over time.
  Active range of motion of the neck, Head repositioning accuracy, hand strength, neck muscle endurance, sharpened Romberg, walking in a figure of eight, neurological examination: reflexes, sensibility and motor function
SF-36 | Baseline and at 3 month follow-up. The outcome measure is going to report a change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, Assoc. Prof., Study Chair — Linkoeping University
Locations (1):
- Anneli Peolsson, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peolsson A, Landen Ludvigsson M, Tigerfors AM, Peterson G. Effects of Neck-Specific Exercises Compared to Waiting List for Individuals With Chronic Whiplash-Associated Disorders: A Prospective, Randomized Controlled Study. Arch Phys Med Rehabil. 2016 Feb;97(2):189-95. doi: 10.1016/j.apmr.2015.10.087. Epub 2015 Oct 26. PMID 26514296
- [Derived] Landen Ludvigsson M, Peterson G, Jull G, Trygg J, Peolsson A. Mechanical properties of the trapezius during scapular elevation in people with chronic whiplash associated disorders--A case-control ultrasound speckle tracking analysis. Man Ther. 2016 Feb;21:177-82. doi: 10.1016/j.math.2015.07.009. Epub 2015 Aug 5. PMID 26277485